CLINICAL TRIAL: NCT06340334
Title: Efficacy and Safety of Tegoprazan Dual Therapy and Furazolidone-based Bismuth Quadruple Therapy for Helicobacter Pylori Eradication: A Prospective, Multicenter, Open-label, Randomized Controlled Clinical Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zhenyu Zhang, Director of Gastroenterology, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20240123-05
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Helicobacter Pylori Infection; Tegoprazan; Furazolidone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): oral Tegoprazan 50 mg, bid+amoxicillin 1000 mg, tid. The duration of treatment is 14 days.
  Interventions: Biological: Tegoprazan-amoxicillin dual therapy
- Group B (Active Comparator): oral Tegoprazan 50 mg, bid + amoxicillin 1000 mg, bid + furazolidone 100 mg, bid + colloidal pectin bismuth 300 mg, bid. The duration of treatment is 14 days.
  Interventions: Biological: Tegoprazan-amoxicillin dual therapy

INTERVENTIONS:
Biological: Tegoprazan-amoxicillin dual therapy — A total of 600 Hp-positive patients who had not received Hp eradication therapy before or had had Hp eradication in the early stage but had not undergone eradication therapy in the past six months were randomly divided into two groups: group A subjects received Tegoprazan 50 mg, bid + amoxicillin 1000 mg, tid; Group B subjects received Tegoprazan 50 mg, bid + amoxicillin 1000 mg, bid + furazolidone 100 mg, bid + colloidal pectin bismuth 300 mg, bid. The duration of treatment is 14 days. The eradication rate, adverse reactions, and compliance of the two groups were compared.
  Other Names: Furazolidone-based Bismuth Quadruple Therapy

SUMMARY:
To compare the efficacy and safety of Tegoprazan-amoxicillin dual therapy and bismuth quadruple therapy based on furazolidone in the treatment of Helicobacter pylori eradication, the eradication rate, patient compliance, and adverse drug reactions of H. pylori infection were compared in a multi-center clinical joint study in Jiangsu Province.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, open-label, randomized, parallel-controlled study. A total of 600 Hp-positive patients who had not received Hp eradication therapy before or who had previously eradicated Hp but had not undergone eradication therapy in the past six months were recruited, and the basic clinical data of the patients (age, gender, drug allergy history, diagnosis and treatment, etc.) were recorded, and they were randomly divided into two groups according to the ratio of 1:1. Group A subjects received oral Tegoprazan 50mg, bid + amoxicillin 1000mg, tid; Group B subjects received oral Tegoprazan 50 mg, bid + amoxicillin 1000 mg, bid + furazolidone 100 mg, bid + colloidal pectin bismuth 300 mg, bid. The duration of treatment is 14 days.

During the 14-day eradication treatment period, all participants were asked to record their adverse reactions and adherence to the medication. On the 7th and 14th days of medication, the researchers will conduct follow-up visits through WeChat or telephone to determine the adverse reactions and compliance of the patients, and observe and record whether the subjects have nausea, diarrhea, dizziness, bitter mouth, rash, constipation and other adverse reactions. In addition, subjects returned to the hospital 4-6 weeks after the end of treatment to check for H. pylori eradication by 13C-UBT or 14C-UBT.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old;
2. Patients who have had a positive 13C or 14C breath test and have not received Helicobacter pylori eradication therapy before, or who have failed to eradicate in the early stage but have not received eradication therapy within half a year;
3. Voluntarily join this trial and sign the informed consent form.

Exclusion Criteria:

1. Allergy to the study drug (penicillin, amoxicillin, furazolidone, Tegoprazan, etc.);
2. Patients with active peptic ulcer disease;
3. Patients who have received Helicobacter pylori eradication therapy within half a year;
4. Use of antibiotics, bismuth, histamine H2 receptor antagonists or PPIs for 4 weeks before starting study treatment;
5. use of adrenocorticosteroids, non-steroidal anti-inflammatory drugs or anticoagulants;
6. History of esophageal or gastric surgery;
7. Pregnant or lactating women;
8. Suffering from serious concomitant diseases, such as liver disease, cardiovascular disease, lung disease, kidney disease;
9. Alcoholism.
10. Gastric mucosa-associated lymphoid tissue lymphoma (MALT), malignant tumor diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | 4-6 weeks after the end of the last dose
  The eradication effect of Helicobacter pylori was detected by 13C-UBT or 14C-UBT

SECONDARY OUTCOMES:
Security observations | Days 7 and 14 of eradication treatment
  Adverse reactions such as nausea, diarrhea, dizziness, change in taste, rash, constipation, etc

OTHER OUTCOMES:
Patient compliance | Within 3 days after the end of treatment
  Actual amount of medication taken as a proportion of the total amount of medication to be taken during the 14-day treatment period

IPD SHARING:
Plan to Share IPD: Yes